CLINICAL TRIAL: NCT03723811
Title: A Multicenter, Placebo Controlled, Randomized, Double Blind, Phase II Study to Evaluate the Efficacy and Safety of SJP002 Eye Drops in Patients With Dry Eye Syndrome.
Brief Title: Clinical Study to Investigate the Efficacy and Safety of SJP002 Ophthalmic Solution in Patients With Dry Eye Syndrome.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Samjin Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SJSJP002_02
Record Dates: First submitted 2018-10-26; First posted 2018-10-30 (Actual); Last update posted 2022-04-07 (Actual); Status verified 2022-03

CONDITIONS: Dry Eye Syndromes
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 1 (Experimental): SJP002 BID
  Interventions: Drug: SJP002 BID
- 2 (Experimental): SJP002 QID
  Interventions: Drug: SJP002 QID
- Placebo 1 (Placebo Comparator): SJP002 Placebo 1
  Interventions: Drug: SJP002 Placebo 1
- Placebo 2 (Placebo Comparator): SJP002 Placebo 2
  Interventions: Drug: SJP002 Placebo 2

INTERVENTIONS:
Drug: SJP002 BID — 1 drop b.i.d for 12 weeks
  Arms: 1
Drug: SJP002 QID — 1 drop q.i.d for 12 weeks
  Arms: 2
Drug: SJP002 Placebo 1 — 1 drop q.i.d for 12 weeks
  Arms: Placebo 1
Drug: SJP002 Placebo 2 — 1 drop q.i.d for 12 weeks
  Arms: Placebo 2

SUMMARY:
This study is to evaluate the efficacy and safety of SJP002 ophthalmic solution compared to placebo in patients with Dry Eye Syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Age over 19.
* Must meet all criteria listed below at least in one eye.

  1. Fluorescein corneal staining score ≥ 2
  2. Schirmer test ≤ 10mm in 5 mins
  3. Tear break-up time ≤ 10 secs

Exclusion Criteria:

* Ocular disorder that may confound interpretation of study results.
* Wearing contact lenses 72 hrs prior to screening visit and unwilling to avoid wearing contact lenses for the duration of the study period.
* History of laser-assisted in situ keratomileusis (LASIK) or similar type of corneal refractive surgery within 12 months prior to screening visit, and/or any other intraocular surgery within 90 days prior to screening visit.
* Female currently pregnant, nursing, or planning a pregnancy; or woman who has a positive pregnancy test.
* Participation in other studies within 30 days of screening visit.

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2017-11-28 (Actual); Primary Completion 2018-06-26 (Actual); Study Completion 2018-06-26 (Actual)

PRIMARY OUTCOMES:
Change from baseline of Fluorescein Corneal Staining(FCS) score | 4 weeks
  The degree of corneal inflammation is scored (total of 5 points) according to the Oxford grading scale from 0 (no staining, A) to 5 (severe, confluent staining, >E).

SECONDARY OUTCOMES:
Change from baseline of Fluorescein Corneal Staining(FCS) score | 2 weeks
  The degree of corneal inflammation is scored (total of 5 points) according to the Oxford grading scale from 0 (no staining, A) to 5 (severe, confluent staining, >E).
Change from baseline of Lissamine Green Conjunctival Staining(LGCS) score | 2, 4 weeks
  Immediately after dyeing (max within 2 minutes), Scored by using slit lamp on white light and a red barrier filte according to the Oxford scheme using a source From 0 (no staining, A) up to 5 (severe, confluent staining, >E) (10 points in total).
Change from baseline of Schirmer Test score | 2, 4 weeks
  Change from Baseline, 2, 4 Weeks
Change from baseline of Tear Break-Up Time(TBUT) | 2, 4 weeks
  Change from Baseline, 2, 4 Weeks
Change from baseline of Standard Patient Evaluation of Eye Dryness questionnaire(SPEED) | 4 weeks
  Change from Baseline, 4 Weeks
Numbers of used artificial tears during the study period | 4 weeks
  Change from Baseline, 4 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Choun-Ki Joo, M.D.,Ph.D., Principal Investigator — Seoul St. Mary's Hospital
Locations (1):
- Seoul St. Mary's Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No